CLINICAL TRIAL: NCT06566703
Title: Testing All Nations Snuff Out Smokeless (ANSOS) for Efficacy in Multi-Tribal Urban Communities
Brief Title: Testing ANSOS for Efficacy in Multi-Tribal Urban Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSG-21-043-01-CPPB
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Smokeless Tobacco Cessation
Keywords: American Indian; smokeless tobacco cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All Nation Snuff Out Smokeless (Experimental): This is a culturally targeted smokeless tobacco cessation program developed for American Indian communities. It includes group sessions via Zoom, individual telephone counseling, and educational materials.
  Interventions: Behavioral: All Nations Snuff Out Smokeless; Behavioral: Healthy Living
- Wait List Control - Healthy Living (Experimental): Participants randomized to this arm are provided with information about healthy living while they wait for their turn at the intervention arm. Participants learn about diet, exercise, and stress reduction. They receive the All Nations Snuff Out Smokeless intervention after a six-month waiting period.
  Interventions: Behavioral: All Nations Snuff Out Smokeless; Behavioral: Healthy Living

INTERVENTIONS:
Behavioral: All Nations Snuff Out Smokeless — All Nations Snuff Out Smokeless is a culturally tailored smokeless tobacco cessation program that incorporates group-based and individual counseling.
Behavioral: Healthy Living — Healthy Living is an educational program that provides information about diet, exercise, stress, and general health. It uses group-based and individual discussion, along with educational materials.

SUMMARY:
This is a wait-list control trial to test for efficacy of the All Nations Snuff Out Smokeless (ANSOS) recreational tobacco cessation program in multi-tribal American Indian (AI) communities. Participants randomized to the control arm are provided with a Healthy Living educational intervention while they wait for the program to encourage them to remain engaged with the study team during the six-month waiting period. Participants from the ANSOS arm are offered the Healthy Living educational intervention after they complete the 6-month outcome measures.

DETAILED DESCRIPTION:
All Nations Snuff Out Smokeless (ANSOS) is a culturally tailored, group-based quit smokeless tobacco (SLT) program for American Indian (AI) people. Intervention components are described below.

Group Support Sessions: The primary component of ANSOS are four group-based support sessions, led by an AI facilitator, conducted via Zoom. All group sessions begin with team building and discussion about things people are experiencing in their lives, both those related directly to recreational tobacco use and other things that help or hinder quit attempts. The first group session is devoted to forming a cohesive group and learning about individual journeys with tobacco. Additional group sessions focus on topics covered in the education curriculum.

Individual Telephone Counseling: After initial group sessions, facilitators call participants weekly to see how they are doing, discuss personal issues related to the quitting process, and to remind them of the next group.

Educational Curriculum: The ANSOS curriculum includes 11 brochures, given throughout the program; it combines cessation information with cultural elements. Topics covered include substantial information about tobacco as a sacred plant for many, though not all, AI tribes, historical trauma, and medical/research mistrust issues, among other topics related to how to effectively quit using recreational tobacco products. Educational materials for this project will be given to participants electronically via pdf documents.

Healthy Living is an educational program primarily designed to maintain the interest of participants in the control arm in continuing into the ANSOS program after their 6-month waiting period. It includes group-based educational discussion about healthy diet, exercise, and stress management, along with educational materials on these topics. Participants also receive individual discussion with program facilitators in between group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Stable telephone number that can be used for the purpose of the study
* Willing to be followed for 12 months and participate in study activities
* Able to attend Zoom sessions
* Current SLT user, at least once per day
* Self-reported AI

Exclusion Criteria:

* Cannot provide a stable phone number for 12 months for the purpose of the study
* Unable to attend Zoom sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 7-day point prevalence abstinence | 6 months
  7-day point prevalence abstinence from smokeless tobacco product use

SECONDARY OUTCOMES:
Number of participants with continuous abstinence | 6 months, 12 months
  Continuous abstinence from smokeless tobacco product use

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Daley, PhD, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No